CLINICAL TRIAL: NCT00866671
Title: A Multicentre, Single Arm, Observational Phase IV Study to Assess the Safety and Efficacy of Nelarabine in Children and Young Adults (up to 21 Years of Age) With Relapsed or Refractory T-Lineage Acute Lymphoblastic Leukaemia or Lymphoblastic Lymphoma
Brief Title: Observational Study of Nelarabine in Children and Young Adults
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111081
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Leukaemia, Lymphoblastic, Acute
Keywords: T-ALL; Safety; Post Authorisation Safety Study; T-LBL; Lymphoblastic Lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — nelarabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nelarabine: nelarabine 650mg/m2 IV daily for 5 days. repeat every 21 days.
  Interventions: Drug: nelarabine

INTERVENTIONS:
Drug: nelarabine — Nelarabine is a prodrug of 9-β-D-arabinofuranosylguanine (ara-G), a deoxyguanosine analogue.

SUMMARY:
This international, multicentre, single arm, phase IV study will assess the safety and efficacy of nelarabine in children and young adults with relapsed or refractory T-lineage acute lymphoblastic leukaemia (T-ALL) or lymphoblastic lymphoma (T-LBL) whose disease has not responded to or has relapsed following treatment with at least two chemotherapy regimens. It is a post-authorisation safety study (PASS) conducted for the purpose of confirming the safety profile and the clinical benefit of nelarabine under licensed conditions of use. The study is observational, non-interventional, and will include approximately 40 children and young adults (up to 21 years of age).

ELIGIBILITY:
Inclusion Criteria:

* ≤ 21 years of age
* Relapsed or refractory T-lineage acute lymphoblastic leukaemia (T-ALL) or lymphoblastic lymphoma (T-LBL)
* Prior treatment with at least two chemotherapy regimens
* Selected for treatment with nelarabine

Exclusion Criteria:

* Known hypersensitivity to the active substance.
* Women of childbearing potential who are unable or unwilling to use adequate contraceptive measures
* Males with partners of child bearing potential who are not willing to use condoms or abstinence
* Patients with persistent neurological toxicity (CTC grade > = grade 2)
* Adolescents (aged 16 years and over) and adults for whom the physician prescribes the 1500mg/m2 dose of nelarabine.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male or Female 21 years or younger with Relapsed or refractory T-lineage Acute Lymphoblastic Leukaemia (T-ALL) or lymphoblastic lymphoma (T-LBL)
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Neurological adverse events | Up to one year after treatment

SECONDARY OUTCOMES:
Other adverse events | Up to one year after treatment
clinical response rate and survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- Denmark (4):
  - GSK Investigational Site, Aahur N
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Koebenhavn Oe
  - GSK Investigational Site, Odense C
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (2):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Essen, North Rhine-Westphalia
- Israel (4):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
- GSK Investigational Site, Bologna, Emilia-Romagna, Italy
- GSK Investigational Site, Rotterdam, Netherlands
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (2):
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Boadilla Del Monte (Madrid)
  - GSK Investigational Site, Madrid